CLINICAL TRIAL: NCT03725280
Title: Micro RNA Profile in the Ovarian Follicle Fluid of Transgender Men Treated With Testosterone and the Association With Fertility Potential
Brief Title: Micro RNA Profile in the Ovarian Follicle Fluid of Transgender Men
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: University of California, San Diego (Other)
Responsible Party: Principal Investigator, michal roll, Research & Development Director, Tel-Aviv Sourasky Medical Center
Other Study IDs: 0645-18
Record Dates: First submitted 2018-10-04; First posted 2018-10-31 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: IVF; Fertility Preservation; Infertility
Keywords: Micro RNA; Ovarian Follicular fluid; Transgender men; Testosterone
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Transgender men I: Transgender men after testosterone treatment
  Interventions: Procedure: IVF
- Transgender men II: Transgender men before testosterone treatment
  Interventions: Procedure: IVF
- IVF- PCOS: IVF- PCOS patients with high testosterone levels
  Interventions: Procedure: IVF
- Egg donors: IVF- egg donors patients
  Interventions: Procedure: IVF

INTERVENTIONS:
Procedure: IVF — None interventional study (Collection of ovarian follicular fluid during IVF treatment)
  Other Names: not interventional study

SUMMARY:
The effects of gender transitioning, particularly the effects of testosterone exposure in transgender men, on the oocyte and embryo development are largely unknown. Based on prior studies suggesting that the extracellular RNAs secreted by the ovarian follicle cells reflect the oocyte and embryo biological state, the investigators propose to use these extracellular RNAs to gain insights into the effects of testosterone exposure in transgender men on their oocyte and embryo without impacting the clinical IVF process.

DETAILED DESCRIPTION:
Background:

MicroRNAs are small RNA molecules that control gene expression in the cell. micro RNAs are also found in the body fluids in vesicles known as exosomes that interact with cellular membranes, release their contents, thus responsible for cell-to-cell contact.

The ovarian follicle fluid contains various substances, including micro RNAs, which are secreted by the various follicle cells and plays an important role in the development and maturation of the oocyte. Recent studies have found that micro RNAs found in the follicle fluid play an important role in the maturation of the oocyte, fertilization, embryo quality, and implantation.

Transgenderism is an umbrella term describing people whose gender identity and/or expression does not align with their sex assigned at birth. A transgender man is a man who was assigned female at birth. The medical interventions for transgender men include hormonal (testosterone) treatment that can negatively affect fertility, and fertility preservation is an option to overcome this potential damage. The fertility preservation options for transmen include oocyte and embryo cryopreservation. The American Society for Reproductive Medicine (ASRM) recommends that: 1. All transgender patients will be counseled regarding the fertility options prior to initiating the medical transition. 2. Transgenders have to preserve gametes (cryopreservation) before starting hormonal therapy. 3. Transgenders that are already using cross-sex hormone treatment have to stop hormone treatment for at least 3 months before fertility preservation. The aim of the current study is to compare the micro RNA profile of the follicle fluid of IVF patients exposed to high testosterone levels with IVF patients with normal testosterone levels and examine the possible association between testosterone exposure and fertility potential.

Specific aims:

1. To characterize the profile of extracellular RNAs in the follicle fluid of transgender patients treated with testosterone.
2. To determine the association of the follicle fluid RNA profile in these patients with the number and quality of oocyte, fertilization potential and the quality of the embryos.

Research plan

Research Location:

IVF Unit, Lis Maternity Hospital, The Tal Aviv Sourasky Medical Center (TASMC) Department of Reproductive Medicine, Division of Maternal Fetal Medicine, University of California, San Diego (UCSD)

Estimated duration: 5 years

Study size: 40 IVF patients: 10 transgender men after testosterone therapy, 10 transgender men before testosterone therapy, 10 patients with the polycystic ovarian syndrome and high endogenic testosterone levels, 10 egg donors

Research design and methods

1. Patients who are intended to participate in the study will receive a detailed explanation of the study and will sign a consent form.
2. IVF patients included in the study will be referred to all tests routinely required prior to IVF procedure, including blood tests for hormonal profile and testosterone levels, and ultrasound for antral follicle count (AFC). Testosterone levels in transgender patients will be tested before and after testosterone therapy is stopped.
3. Patients will get an IVF protocol including hormonal therapy which will be followed by the oocyte retrieval.
4. During oocyte retrieval, follicular fluids will be collected from IVF cycles of 10 transgender patients exposed to testosterone and 30 control patients not exposed to external testosterone (10 transgender men before testosterone therapy, 10 patients with the polycystic ovarian syndrome and high endogenic testosterone levels, 10 egg donors). These biofluids will be discarded materials obtained during the course of clinical IVF cycles.

   The samples of the follicular fluid will be subjected to unrecognized samples with a running number, encoded, thus eliminating any possibility of establishing contact with the particular patient.
5. The follicular fluid will undergo centrifugation and the supernatant will be maintained at -80 degrees in the IVF unit, TASMC.
6. Follicular fluid from clinical IVF cycles from enrolled transgender subjects and controls, along with non-identifiable patient information associated with each follicular fluid and embryo culture fluid sample, including patient age, BMI, use of testosterone, cause of IVF treatment, number of oocytes, number of fertilized oocytes and the quality of embryos, will be transferred from the Amir group at TASMC to the Laurent group at UCSD.
7. At UCSD, extracellular RNA will be isolated from the follicle fluid samples using The Norgen and The ExoRNeasy methods (followed by qRT-PCR validation) and subjected to RNA sequencing analysis using NEBNext multiple small RNAseq library preparation kits.
8. The resulting RNAseq data will be analyzed to identify changes in micro RNA expression associated with clinical variables, including the cause of IVF, testosterone treatment, and embryo quality.

Steps 1-6, 8 will be performed in TASMC. Steps 7-8 will be performed in UCSD.

Inclusion criteria:

* Patients aged 18 and older

Exclusion criteria:

* Patients under 18 years old
* Patients who did not respond to hormone therapy and the IVF cycle was discontinued.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and older.

Exclusion Criteria:

* Patients under 18 years old.
* Patients who did not respond to hormone therapy and the IVF cycle was discontinued.

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Female undergoing IVF treatments for fertility preservation/infertility/egg donation
Study Population: Transgender men before testosterone therapy Transgender men after testosterone therapy, Patients with polycystic ovarian syndrome (PCOS) and high testosterone levels undergoing IVF treatments Egg donors undergoing IVF treatments
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Characterization of micro RNA profile in follicle fluid of transgender men treated with testosterone. | 5 years
  The follicle fluid of transgender men will be collected during egg retrieval, and micro RNA will be isolated from the follicle fluid samples using The Norgen and The ExoRNeasy methods (followed by qRT-PCR validation) and subjected to RNA sequencing analysis using NEBNext multiple small RNAseq library preparation kits. Total Testosterone levels (ng/ml) in the blood will be examined in all patients prior to the IVF treatment.

SECONDARY OUTCOMES:
The association between micro RNA profile in follicle fluid of transgender men and the number of eggs. | 5 years
  Expert embryologists will count the eggs after egg retrieval and the number of the eggs will be correlated to the micro RNA profile from the follicle fluid of transgender men.
The association between micro RNA profile in follicle fluid of transgender men and the maturation level of the eggs. | 5 years
  Eggs will be denuded immediately after egg collection and the in vivo egg M-Index will be calculated for the egg cohort collected (number of normal metaphase II eggs per total number of normal eggs which will be collected), and the M-index will be correlated to the micro RNA profile from the follicle fluid of transgender men.
The association between micro RNA profile in follicle fluid of transgender men and the embryo quality. | 5 years
  Blastocyst quality will be evaluated according to Gardner's scoring system and three subgroups will be classified: high (blastocysts or hatched blastocysts with inner cell mass [ICM] and trophectoderm morphology of grade AA/AB/BA), low (delayed embryos at <9 cells or blastocysts with ICM or trophectoderm morphology of grade C), and moderate (all of the rest). The embryo quality will be correlated to the micro RNA profile from the follicle fluid of transgender men.
The association between micro RNA profile in follicle fluid of transgender men and the embryo development level. | 5 years
  All embryos will be incubated in the integrated EmbryoScopeTM time-lapse monitoring system (EmbryoScopeTM; Vitrolife, Sweden) and morphkinetic parameters will be analyzed by time-lapse technology on days 1-5. The embryo developmental level will be correlated to the micro RNA profile from the follicle fluid of transgender men.

IPD SHARING:
Plan to Share IPD: No